CLINICAL TRIAL: NCT04458038
Title: Does Chronic Obstructive Lung Disease Influence the Cognitive Function: Assessment Using a Driving Simulator and Other Cognitive Tests
Brief Title: Does Chronic Obstructive Lung Disease Influence the Cognitive Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sygehus Lillebaelt (Other)
Collaborators: Chiesi Foundation (Unknown); Overlæge Jørgen Werner Schous og hustru, Else-Marie Schou, født Wonge´s Fond (Unknown); Danmarks Lungeforening (Other)
Responsible Party: Principal Investigator, Kristina Kock Hansen, Master of Science in Health Science, Sygehus Lillebaelt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19/44919
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention arm (Experimental)
  Interventions: Other: driving simulator

INTERVENTIONS:
Other: driving simulator — For this study a driving simulator is being used which is an internationally approved method. Besides the driving simulator following tests are done: COPD Assessment Test (CAT), Hospital Anxiety and Depression Scale (HADS), Montreal Cognitive Assessment (MoCA), a clock drawing test and a continuous reaction time test (CRT). A CardioRespiratory Monitor (CRM), NOX T3TM, is used to measure if the patients have moderate to severe OSA. Furthermore, following tests are done: Epworth Sleepiness Scale (ESS).
  Other Names: continuous reaction time test (CRT); cardiorespiratory monitor (CRM)

SUMMARY:
Studies have documented impaired cognitive function in patients with COPD. The possible reasons for this and correlation to the severity of the disease are not well described. This explorative study examines the cognitive skills of COPD patients, quantified by their ability to drive a vehicle and other cognitive test. Furthermore, we want to study the cognitive skills in COPD patients before and after they are diagnosed with and treated for obstructive sleep apnoea (OSA). The overall hypothesis is that chronic lung patients´ cognitive skills correlate with the severity of their disease. We expect that their ability to drive a vehicle drops in relation to the severity of the disease and to comorbidities.

DETAILED DESCRIPTION:
200 COPD patients recruited from the outpatient clinic at the Department of Respiratory Diseases at Vejle Hospital. Approximately 2600 COPD patients are treated in Vejle.

For this study a driving simulator is being used. The subjects are placed in front of a computer monitor which simulates a horizon on the middle of the screen, and a road that appears in the bottom half of the screen. The subjects are encouraged to keep the virtual vehicle on the road, using a steering wheel in front of them. Simultaneous, they are required to keep focus on both sides of the screen where a line of numbers is frequently changing. Every time the number 2 occurs, the subjects must press a button on the steering wheel.

The subjects´ overall ability to control the driving simulator is being expressed by the standard deviation (sd) of distance of the car´s centre to the centre of the road and the number of off-road events. Relevant cognitive measurements, such as reaction speed and ability to split attention, are quantified by the reaction speed to the occurrence of the number 2. The reason for this is that the software of the simulator measures the mean reaction time from the number have occurred until the correct button is pressed, and the number of nil-responses, where the number 2 is not detected.

Every participating subject will receive a 5 minutes testing period of the simulator followed by 30 minutes of applicable driving time.The other tests will be performed/collected just after the driving test.

Besides the driving simulator and tests (see sections below) following are obtained: 1) Lung function (FEV1, FVC and FEV1/FVC), 2) Arterial blood sample including PaO2, PaCO2 and carbonmonooxidhemoglobin (HbCO) (1.5 ml), 3) Smoking status and number of pack years, 4) Status of oxygen therapy, 5) Number of COPD exacerbations in the last year, 6) Comorbidities such as diabetes, metabolic diseases, cardiovascular diseases, kidney insufficiency, 7) Medicine, 8) Height and weight, 9) Level of education, 10) Degree of dyspnoea Medical research Council breathlessness scale (MRC-scale) and 11) Global initiative for chronic Obstructive Lung Disease (GOLD) classification of airflow limitation.

The blood samples will be analysed immediately after they are taken, and as a consequence no biobank will be established. The information will be gathered from the journals and from patient interview in connection with the trial. The information will be used in the assessment of possible reasons to COPD patients´ expected reduced cognitive skills.

The NOX T3TM (see section below) will be delivered in connection with the trial. If the patients are diagnosed with OSA they will shortly after receive standard treatment in the public Sleep Clinic at Vejle Hospital, if the patients accept. After 2-3 month of treatment, the patients will repeat all the tests and blood samples, except the cardiorespiratory monitoring.

To exclude that an improvement of skills is not due to the patients having learned how to improve the test, we will establish a control group. The control group must consist of COPD patients without OSA who must perform a retest like the patients with OSA.

ELIGIBILITY:
Inclusion Criteria:

1. Doctor-diagnosed chronic obstructive lung disease (forced expiratory volume in the first second (FEV1) / forced expiratory vital capacity (FVC) <0.70).
2. Severity of COPD - GOLD 3+4 (GOLD 2019 classification).
3. No exacerbations in the last 6 weeks (aggravation of the respiratory symptoms compared with habitual state, which require treatment).
4. Age ≥ 40 years and ≤ 75 years
5. The patient must have driven a vehicle within the last 3 months.

Exclusion Criteria:

1. Lacking the ability to operate the driving simulator (physical deformities or lack of comprehensive skills to understand instruction of operating the simulator).
2. No valid driver´s license.
3. Do not read and understand Danish.
4. Known obstructive sleep apnoea (OSA).
5. Alcohol consumption (>21 units per week for men, >14 units per week for women).
6. Consumption of alcohol and/or narcotics within the last 24 hours.
7. Uncorrected sight- or hearing reduction.
8. Unstable ischemic heart disease, uncontrolled hypertension or diabetes, left sided heart failure, serious neurologic conditions, cancer, phlebitis, severe psychiatric diseases, uncontrolled thyroid disease or former apoplexy.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Standard deviation from center of the road and number of off-road events | 3 years
  driving simulator

CONTACTS AND LOCATIONS:
Locations (1):
- Sygehus Lillebaelt, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hansen KK, Lokke A, Jensen HI, Gantzhorn EK, Farver-Vestergaard I, Hilberg O. Examining the impact of obstructive sleep apnea on cognitive function in severe COPD. Sleep Breath. 2024 Dec 14;29(1):59. doi: 10.1007/s11325-024-03228-5. PMID 39673053